CLINICAL TRIAL: NCT05670275
Title: Microecology and Host Immunity in Patients With Severe COVID-19 Infection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, wang kaifei, Chinese PLA General Hospital, Chinese PLA General Hospital
Other Study IDs: Respiratory microecology
Record Dates: First submitted 2023-01-02; First posted 2023-01-04 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Microbiome,Immune Function, Critically Ill
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — bronchoalveolar lavage specimens
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study was to analyze the relationship between the microbial community, host immunity and the prognosis of patients with severe COVID-19.

DETAILED DESCRIPTION:
Methods: Bronchoalveolar lavage specimens of patients with severe COVID-19 were collected and studied to analyze the relationship between the composition of patients' microecology and the occurrence and development of disease.

ELIGIBILITY:
Inclusion Criteria:

* 1) Respiratory distress, respiratory rate ≥ 30 times/minute

  2) At rest, oxygen saturation ≤ 93%

  3）PaO2/FiO2 ≤300mmHg

  4) Shock

  5) Respiratory failure requires mechanical ventilation

  6) Complicated with other organ failure requires ICU monitoring and treatment

  7) Or in case of any of the following conditions, even if none of the above conditions is found, it is also managed as a critical case: ① pulmonary imaging shows that the lesion has significantly progressed more than 50% within 24-48 hours; ② Age>60 years old; ③ Complicated with serious chronic diseases (including diabetes, hypertension, coronary heart disease, malignant tumor, structural lung disease, pulmonary heart disease and immunosuppressed population)

Exclusion Criteria:

* 1) Pregnant women

  2) Age<18

  3) Mental disorders

  4) Patients with long-term mechanical ventilation for more than 60 days

  5) Disagreement group researcher

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with severe COVID-19 infection after endotracheal intubation
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
death | 28 day
  mortality

CONTACTS AND LOCATIONS:
Locations (1):
- PLA, Beijing, Beijign, China